CLINICAL TRIAL: NCT04369703
Title: Copeptin as a Biomarker for Central Diabetes Insipidus Development Following Pituitary Surgery
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Dana Erickson, Associate Professor of Medicine, Mayo Clinic
Other Study IDs: 19-010785
Record Dates: First submitted 2020-03-02; First posted 2020-04-30 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Sellar and Suprasellar Masses; Pituitary Tumor
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Access the optimal cut point value of copeptin which predicts development of central diabetes insipidus postoperatively with highest accuracy.
2. Access the optimal cut point value of copeptin which predicts the lack of central diabetes insipidus postoperatively with highest accuracy
3. Access the relative change in copeptin values between baseline and post-surgery as a predictor for diabetes insipidus development.

DETAILED DESCRIPTION:
Patient serum levels of copeptin would be measured after phlebotomy of 3 ml of blood in EDTA tube twice a) within 1-4 hours of extubation and b) within 4-24 hours of extubation (the morning following surgery).

ELIGIBILITY:
Inclusion Criteria:

* Patients with sellar and suprasellar masses who undergo neurosurgical procedure at Mayo Clinic Rochester.

Exclusion Criteria:

* Patients with preexisting CDI.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sellar and suprasellar masses.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Predict central diabetes insipidus development | 2 years
  Using the measured lab value, we will access the optimal cut point value of copeptin which predicts development of central diabetes insipidus postoperatively with highest accuracy.
Predict lack of central diabetes insipidus development | 2 years
  Using the measured lab value, we will access the optimal cut point value of copeptin which predicts the lack of central diabetes insipidus postoperatively with highest accuracy
Assess relative change | 2 years
  Using the measured lab value, we will access the relative change in copeptin values between baseline and post-surgery as a predictor for diabetes insipidus development.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Erickson, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials